CLINICAL TRIAL: NCT05227872
Title: Dynamic Changes in Portal Vein Flow in Decongestion of Patients With Heart Failure and Cardio-Renal Syndrome
Brief Title: PVF in Decongestion of Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, Principal Investigator, Assiut University
Other Study IDs: DCPVFDPHF
Record Dates: First submitted 2021-10-29; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decompensated HF
  Interventions: Device: ultrasound
- Compensated HF
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — POCUS

SUMMARY:
Evaluate PVF alterations in patients with ADHF at arrival and after decongestive treatment

DETAILED DESCRIPTION:
Hospitalizations from heart failure have been shown to be preceded by a gradual increase in cardiac filling pressures using invasive ambulatory monitoring measurements [1, 2]., this technique does not directly assess congestion. The use of point-of-care ultrasound (POCUS) to evaluate lung congestion has been shown to decrease decompensations and urgent heart failure visits [3, 4]. However, besides lung congestion, the abdominal compartment contributes significantly to deranged cardiac as well as renal function in congestive heart failure (CHF) [5].There is increasing recognition that worsening renal function in CHF is related to altered renal blood flow [6, 7]. Recently, alterations in renal venous flow (IRVF) assessed by Doppler imaging have been associated with worse outcomes in patients with CHF [8, 9]. Besides IRVF alterations, portal vein flow (PVF) alterations have been proposed as a marker of venous congestion and right ventricular dysfunction [10, 11]. PVF and IRVF alterations have been shown to correlate with each other and were independently associated with the development of subsequent acute kidney injury (AKI) in patients undergoing cardiac surgery [12, 13]. Portal vein (PV) Doppler is easily obtainable and less time consuming than intra renal venous Doppler. Given the potential usefulness of evaluating venous congestion via POCUS of PVF, we decided to study the dynamic changes that occur during decongestion in patients presenting with heart failure to the emergency department Optimal method for noninvasive assessment of venous congestion remains an unresolved issue. Portal vein (PV) and intra renal venous flow alterations are markers of abdominal venous congestion and have been associated with acute kidney injury (AKI) in cardiac surgery patients. It is currently unknown if portal vein flow (PVF) alterations in heart failure can be reversed with diuretic treatment and track decongestion

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Patients presented with acute decompensated heart failure (either de novo HF or chronic decompensated HF) fulfilling the following criteria: new or worsening HF symptoms (including dyspnea, decreased exercise capacity, fatigue, or other volume overload symptoms), physical examination findings compatible with HF (peripheral edema, pulmonary congestion, increased jugular venous pressure or third heart sound)

Exclusion Criteria:

1. age below 18.
2. pregnant.
3. cardiogenic shock, or hemodynamic instability.
4. Patients with previously diagnosed Child-Pugh B or C liver cirrhosis, liver transplant, or ESRD on renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross-sectonal
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Portal vein in mm in patients with acute decmpensated heart failure | Baseline
  determine the portal vein flow alteration in mm in patients with acute decompensated heart failure and in patients with cardio renal syndrome

SECONDARY OUTCOMES:
Differences in portal vein flow in mm in patients with acute decompensated heart failure and compensated HF in cardiorenal syndrome | Baseline
  Determine the differences between portal vein flow in mm in patients with acute decmpensated heart failure and those with compensated heart failure in patients with cardio renal syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Ellison DH. Why Are Physicians So Confused about Acute Heart Failure? N Engl J Med. 2019 Dec 12;381(24):2374-2375. doi: 10.1056/NEJMc1913976. No abstract available. PMID 31826353
- [Background] Arrigo M, Jessup M, Mullens W, Reza N, Shah AM, Sliwa K, Mebazaa A. Acute heart failure. Nat Rev Dis Primers. 2020 Mar 5;6(1):16. doi: 10.1038/s41572-020-0151-7. PMID 32139695
- [Background] Rivas-Lasarte M, Alvarez-Garcia J, Fernandez-Martinez J, Maestro A, Lopez-Lopez L, Sole-Gonzalez E, Pirla MJ, Mesado N, Mirabet S, Fluvia P, Brossa V, Sionis A, Roig E, Cinca J. Lung ultrasound-guided treatment in ambulatory patients with heart failure: a randomized controlled clinical trial (LUS-HF study). Eur J Heart Fail. 2019 Dec;21(12):1605-1613. doi: 10.1002/ejhf.1604. Epub 2019 Oct 31. PMID 31667987
- [Background] Araiza-Garaygordobil D, Gopar-Nieto R, Martinez-Amezcua P, Cabello-Lopez A, Alanis-Estrada G, Luna-Herbert A, Gonzalez-Pacheco H, Paredes-Paucar CP, Sierra-Lara MD, Briseno-De la Cruz JL, Rodriguez-Zanella H, Martinez-Rios MA, Arias-Mendoza A. A randomized controlled trial of lung ultrasound-guided therapy in heart failure (CLUSTER-HF study). Am Heart J. 2020 Sep;227:31-39. doi: 10.1016/j.ahj.2020.06.003. Epub 2020 Jun 15. PMID 32668323
- [Background] Abu-Saleh N, Aronson D, Khamaisi M, Khoury EE, Awad H, Kabala A, Ramadan R, Karram T, Kakiashvili E, Bishara B, Abassi Z. Increased Intra-abdominal Pressure Induces Acute Kidney Injury in an Experimental Model of Congestive Heart Failure. J Card Fail. 2019 Jun;25(6):468-478. doi: 10.1016/j.cardfail.2019.03.008. Epub 2019 Mar 14. PMID 30880249
- [Background] Mentz RJ, O'Connor CM. Pathophysiology and clinical evaluation of acute heart failure. Nat Rev Cardiol. 2016 Jan;13(1):28-35. doi: 10.1038/nrcardio.2015.134. Epub 2015 Sep 15. PMID 26370473
- [Background] Tang WH, Kitai T. Intrarenal Venous Flow: A Window Into the Congestive Kidney Failure Phenotype of Heart Failure? JACC Heart Fail. 2016 Aug;4(8):683-6. doi: 10.1016/j.jchf.2016.05.009. Epub 2016 Jul 6. No abstract available. PMID 27395345
- [Background] Iida N, Seo Y, Sai S, Machino-Ohtsuka T, Yamamoto M, Ishizu T, Kawakami Y, Aonuma K. Clinical Implications of Intrarenal Hemodynamic Evaluation by Doppler Ultrasonography in Heart Failure. JACC Heart Fail. 2016 Aug;4(8):674-82. doi: 10.1016/j.jchf.2016.03.016. Epub 2016 May 11. PMID 27179835
- [Background] Husain-Syed F, Birk HW, Ronco C, Schormann T, Tello K, Richter MJ, Wilhelm J, Sommer N, Steyerberg E, Bauer P, Walmrath HD, Seeger W, McCullough PA, Gall H, Ghofrani HA. Doppler-Derived Renal Venous Stasis Index in the Prognosis of Right Heart Failure. J Am Heart Assoc. 2019 Nov 5;8(21):e013584. doi: 10.1161/JAHA.119.013584. Epub 2019 Oct 19. PMID 31630601
- [Background] Eljaiek R, Cavayas YA, Rodrigue E, Desjardins G, Lamarche Y, Toupin F, Denault AY, Beaubien-Souligny W. High postoperative portal venous flow pulsatility indicates right ventricular dysfunction and predicts complications in cardiac surgery patients. Br J Anaesth. 2019 Feb;122(2):206-214. doi: 10.1016/j.bja.2018.09.028. Epub 2018 Nov 28. PMID 30686306
- [Background] Singh NG, Kumar KN, Nagaraja PS, Manjunatha N. Portal venous pulsatility fraction, a novel transesophageal echocardiographic marker for right ventricular dysfunction in cardiac surgical patients. Ann Card Anaesth. 2020 Jan-Mar;23(1):39-42. doi: 10.4103/aca.ACA_250_18. PMID 31929245
- [Background] Beaubien-Souligny W, Benkreira A, Robillard P, Bouabdallaoui N, Chasse M, Desjardins G, Lamarche Y, White M, Bouchard J, Denault A. Alterations in Portal Vein Flow and Intrarenal Venous Flow Are Associated With Acute Kidney Injury After Cardiac Surgery: A Prospective Observational Cohort Study. J Am Heart Assoc. 2018 Oct 2;7(19):e009961. doi: 10.1161/JAHA.118.009961. PMID 30371304
- [Background] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297